CLINICAL TRIAL: NCT07310225
Title: The Effect of the Mediterranean Diet on Metabolic Parameters in Individuals With Type 2 Diabetes: A Comparative Evaluation With the DASH and MIND Diets
Brief Title: Mediterranean Diet vs DASH and MIND in T2DM
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Nurefşan KONYALIGİL ÖZTÜRK, Assist. Prof. Dr, Abant Izzet Baysal University
Other Study IDs: AIBU-BD-NKÖ-03
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes
Keywords: Mediterranean diet; DASH diet; MIND diet
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with Type 2 diabetes: This cohort includes adult participants diagnosed with Type 2 diabetes. No control group is included.
  Interventions: Other: No intervention (observational study)

INTERVENTIONS:
Other: No intervention (observational study) — No intervention (observational study)

SUMMARY:
In our study, we aimed to comparatively evaluate the relative effects of the Mediterranean, DASH, and MIND diets on metabolic parameters in individuals with type 2 diabetes. The study was conducted on 90 individuals diagnosed with T2DM according to the American Diabetes Association diagnostic criteria (fasting blood glucose ≥ 126 mg/dL, 2-hour blood glucose ≥ 200 mg/dL during an oral glucose tolerance test (OGTT), or HbA1c ≥ 6.5% (48 mmol/mol)). Volunteers who participated in the study completed a questionnaire form that included sociodemographic characteristics. In addition, participants' anthropometric measurements (body weight (BW), height, waist circumference (WC), hip circumference (HC), body mass index (BMI)), biochemical parameters (fasting blood glucose, hbA1c (%), LDL-cholesterol, triglycerides, total cholesterol), Visceral Adiposity Index (VAİ), body composition analyses (Fat Mass (FM (%), Fat-Free Mass (FFM) (kg), Basal Metabolic Rate (BMR) (kcal), Visceral Fat Area (VFA) (%)), nutritional status (food consumption frequency, food consumption record, Mediterranean Diet Scale, DASH diet adherence score, and MIND diet adherence score) were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over 19 years of age
* Individuals who are literate
* Individuals diagnosed with Type 2 diabetes

Exclusion Criteria:

* Individuals who have had an acute infection or inflammatory disease within the past month
* Individuals with chronic infectious or inflammatory diseases
* Individuals with cancer

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was designed as a cross-sectional descriptive study. The study included patients who presented to the Internal Medicine Outpatient Clinic at BAİBÜ İzzet Baysal Education and Research Hospital and diagnosed with T2DM according to the American Diabetes Association diagnostic criteria (fasting blood glucose ≥ 126 mg/dL, 2-hour blood glucose ≥ 200 mg/dL during an oral glucose tolerance test (OGTT), or HbA1c ≥ 6.5% (48 mmol/mol)).
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Questionnaire Form | 9 months
  Sociodemographic characteristics of the individuals (age, gender, smoking and alcohol use) were questioned.
Body Weight (BW) | 9 months
  BW was measured using a calibrated digital scale placed on a flat, tiled surface. The scale was sensitive to 100 grams.
Height | 9 months
  Height was measured using a stadiometer with the participant's head positioned in the Frankfort plane and feet placed together.
Waist Circumference (WC) | 9 months
  WC was measured at the midpoint between the lowest rib and the iliac crest (cristal point) using a flexible measuring tape.
Hip Circumference (HC) | 9 months
  HC was measured at the widest point of the hips using a flexible measuring tape.
Body Mass Index (BMI) | 9 months
  BMI was calculated by dividing body weight (in kilograms) by the square of height (in meters): BMI = weight (kg) / height² (m²).
Fasting Blood Glucose | 9 months
  Fasting blood glucose was measured using standard laboratory techniques during routine outpatient visits.
Triglycerides | 9 months
  Triglyceride levels were measured via fasting blood samples analyzed in the outpatient clinic laboratory.
LDL-Cholesterol | 9 months
  LDL-cholesterol was measured from fasting serum samples using standard enzymatic colorimetric methods.
Total Cholesterol | 9 months
  Total cholesterol was measured using routine biochemical analysis in a certified laboratory.
HbA1c (%) | 9 months
  Fasting blood glucose was measured using standard laboratory techniques during routine outpatient visits.
Abdominal obesity index (VAI) | 9 months
  Abdominal obesity index (VAI): VAI has been used to assess abdominal obesity. VAI (Men) = [Waist circumference (cm) / (36.58 + (1.88 × BMI)] × (triglycerides / 1.03) × (1.31 / HDL-C) , VAI (Women) = [Waist circumference (cm) / (36.58 + (1.88 × BMI)] × (triglycerides / 0.81) × (1.52 / HDL-C)
Body Fat Mass (FM) (%) | 9 months
  Obtained using a bioelectrical impedance analysis (BIA) device (Tanita Innerscan BC 401, Japan).
Basal Metabolic Rate (BMR) (kcal) | 9 months
  Bioelectrical impedance analysis (BIA) device (Tanita Innerscan BC 401, Japan) was used.
Fat-Free Mass (FFM) (kg) | 9 months
  bioelectrical impedance analysis (BIA) device (Tanita Innerscan BC 401, Japan).
Visceral Fat Area (VFA) (%) | 9 months
  Bioelectrical impedance analysis (BIA) device (Tanita Innerscan BC 401, Japan).
Food consumption frequency | 9 months
  Participants were asked about the foods they consumed in the past month from seven groups, including five basic food groups (meat and meat products, milk and dairy products, bread and grains, vegetables and fruits, sugars and fats), beverages, and fast food. Participants were asked how often and in what quantities they consumed these foods using eight options: "every meal," "every day," "5-6 days a week," "3-4 days a week," "1-2 days a week," "once every 15 days," "once a month," and "never." In evaluating food consumption records, responses regarding food consumption frequency were calculated using food consumption frequency. The amounts of food and beverages consumed were multiplied by "3" for "every meal," '1' for "every day," "0.7855" for "5-6 times a week," "0.498" for "3-4 times a week," "0.2145" for "1-2 times a week," "0.067" for "once every 15 days," and "0.033" for "once a month" to obtain the daily average amounts.
Food consumption record | 9 months
  A single-day food consumption record was obtained using the 24-hour recall method to determine participants' food consumption patterns. The Food and Nutrition Photo Catalog was used to estimate portions to ensure that the amounts of food consumed were assessed accurately and reliably. Based on these records, daily energy and nutrient intakes were calculated using the Nutrition Information System (BEBİS) software, based on the type and amount of food consumed by individuals in the last 24 hours.
DASH diet compliance | 9 months
  Individuals' DASH diet compliance scores were calculated based on their food consumption frequency after their energy requirements were calculated. The highest possible score on the DASH diet compliance scale is 8.0. A score of 4.5 or above is considered 'high compliance', while a score below 4.5 is considered 'low compliance'.
Mediterranean diet adherence scale | 9 months
  The Mediterranean Diet Scale was used to determine individuals' adherence to the Mediterranean diet. This scale consists of a total of 14 questions, 2 of which relate to food consumption habits and 12 of which relate to food consumption frequency. Each question is scored as either 0 or 1 point. The scale's scoring range is set at 0-14 points.
MIND diet compliance score | 9 months
  It includes a total of 15 different food groups, consisting of ten groups that protect brain health and five groups that harm brain health. Individuals' food consumption records and frequency of food consumption were examined, and the consumption amounts of foods belonging to these 15 groups were divided into portions and evaluated according to the scoring system. This scale is scored from 0 to 15, and there is no cutoff point for determining compliance with the MIND diet.

CONTACTS AND LOCATIONS:
Locations (1):
- Bolu Abant İzzet Baysal University, Faculty of Health Sciences, Bolu, Turkey (Türkiye)